CLINICAL TRIAL: NCT06942754
Title: Bracing and Reconstruction of the Anterior Cruciate Ligament for Efficacy Trial (BRACE-trial)
Brief Title: Bracing and Reconstruction of the Anterior Cruciate Ligament for Efficacy Trial
Acronym: BRACE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00123098
Record Dates: First submitted 2025-04-16; First posted 2025-04-24 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-04

CONDITIONS: Anterior Cruciate Ligament Injuries
Keywords: Anterior Cruciate Ligament (ACL) reconstruction; postoperative bracing; functional bracing
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Intervention Model Description: A total of 96 patients will be randomized, which means 48 patients will be in the bracing group and 48 in the non-bracing group, based on a sample size calculation. Patients will be randomized during their 2-week post-op visit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- With postoperative brace (DonJoy Defiance Pro) (Experimental): Quadriceps Autograft ACL Reconstruction with the use of post-surgical functional bracing, using the DonJoy Defiance Pro brace
  Interventions: Device: post-surgical functional bracing
- Without post-surgical functional bracing (No Intervention): Quadriceps Autograft ACL Reconstruction without the use of post-surgical functional bracing

INTERVENTIONS:
Device: post-surgical functional bracing — Quadriceps Autograft ACL Reconstruction with the use of post-surgical functional bracing, using the DonJoy Defiance Pro brace
  Other Names: DonJoy Defiance Pro brace
  Arms: With postoperative brace (DonJoy Defiance Pro)

SUMMARY:
Several attempts have been made to reduce these failure rates and improve return to sports rates in high-risk populations, and one of these approaches has been postoperative bracing. A recent survey of the Anterior cruciate ligament (ACL) Study Group has shown that 53% of surgeons prefers functional bracing following ACL reconstruction. Currently, however, there is no clear consensus on whether functional bracing following ACL reconstruction leads to lower failure rates, improved stability or better patient-reported outcomes when compared to ACL reconstruction without bracing.

DETAILED DESCRIPTION:
Given the increased popularity in quadriceps tendon graft, the biomechanical advantages of postoperative functional bracing, and the graft elongation that occurs predominantly with soft tissue grafts, there might be a role for functional bracing following quadriceps ACL reconstruction. Additionally, no studies to date have assessed the role of psychological readiness of return to sport, kinesiophobia and return to sport rates with and without functional bracing following ACL reconstruction (ACLR).

The purpose of this randomized controlled trial is to assess the 2-year outcomes of psychological readiness, patient-reported outcome measures (PROMs), clinical stability, return to sport and failure rates following quadriceps autograft ACL reconstruction with and without functional bracing in the postoperative phase in younger athletic patients and military patients with a higher risk of failure or not returning to sports or duty, respectively, in a randomized study: the Bracing and Reconstruction of the Anterior Cruciate Ligament for Efficacy trial (BRACE-trial).

ELIGIBILITY:
Inclusion Criteria:

* patients with unilateral complete ACL injury
* patients involved in sports and the desire to return to sports
* patients undergoing quadriceps autograft ACL reconstruction
* must be 14 to 39 years old

Exclusion Criteria:

* multiligamentous knee injuries defined as two ligaments requiring surgical stabilization
* concomitant suture tape augmentation, extra-articular tenodesis or anterolateral ligament reconstruction
* concomitant femoral, tibial, or patellar fracture(s)
* patients with significant osteoarthritis
* concomitant ipsilateral knee dislocation or patellar dislocation
* significant lower leg malalignment requiring correcting osteotomies
* prior ACL surgery, including contralateral knee
* pregnancy during injury or surgery
* unable to provide consent
* prolonged use of prednisolone or cytostatics
* comorbidities (e.g., muscular, neurological, vascular) that influence rehabilitation

Ages: 14 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-09-11 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Change in ACL-return to sport index (ACL-RSI) Scores | Baseline and 3, 6, 12, and 24 months
  The ACL-Return to Sport after Injury scale (ACL-RSI) is a 12-item survey that measures psychological readiness to return to sport after an ACL injury or surgery. It uses a visual analog scale from 0 to 100, where higher scores indicate greater psychological readiness. The total score is calculated as a percentage of the 12-item total score.
  A higher ACL-RSI score indicates a greater level of psychological readiness for returning to sport.

SECONDARY OUTCOMES:
Tampa Scale Kinesiophobia 11 (TSK-11) Score | Baseline and 3, 6, 12, and 24 months
  The TSK-11 (Tampa Scale for Kinesiophobia) is a 11-item questionnaire assessing fear of movement/re-injury, scored on a 4-point Likert scale (1-4) with a total score range of 11-44, where higher scores indicate greater fear of pain and movement.
  Lower scores (closer to 11): Indicate minimal or no kinesiophobia (fear of movement/re-injury).
  Higher scores (closer to 44): Suggest a greater degree of kinesiophobia.
International Knee Documentation Committee (IKDC) Score | Baseline and 3, 6, 12, and 24 months
  The IKDC is a patient-completed tool, which contains sections on knee symptoms (7 items), function (2 items), and sports activities (2 items). Scores range from 0 points (lowest level of function or highest level of symptoms) to 100 points (highest level of function and lowest level of symptoms)
Lysholm score | Baseline and 3, 6, 12, and 24 months
  The Lysholm Knee Scoring Scale is a 100-point questionnaire used to assess knee function and is often used to evaluate knee injuries and surgeries, with higher scores indicating better function and fewer symptoms.
  A higher score indicates better knee function and fewer symptoms. Scores are often categorized as excellent (95-100), good (84-94), fair (65-83), and poor (<65).
Forgotten Joint Score (FJS-12) | Baseline and 3, 6, 12, and 24 months
  The Forgotten Joint Score (FJS-12) is a patient-reported outcome measure designed to assess how much a patient is aware of their artificial join in everyday life, with higher scores indicating less awareness and better surgical outcomes.
  Each response is assigned a score (0-4), and the scores are summed and transformed to a 0-100 scale, with higher scores indicating less awareness of the joint.
  Interpretation:
  A higher score suggests that the patient is less aware of their joint, indicating a better outcome and higher satisfaction with the surgery.
SANE Score | Baseline and 3, 6, 12, and 24 months
  The SANE score asks the patient to rate the shoulder on a scale from 0 to 100, with 100 being the patient's normal. Although singular in nature, the SANE score incorporates broad intangible differences in patient-perceived function, quality of life, and goals.
  SANE scores range from 40% to 60% at baseline for most patients before treatment and range from 75% to 85% at 1 year after therapy depending on the condition
5-point Likert Scale for Surgery Satisfaction Score | Baseline and 3, 6, 12, and 24 months
  A 5-point Likert scale for surgery satisfaction typically uses a range from "Very Unsatisfied" to "Very Satisfied" with options like "Very Dissatisfied," "Dissatisfied," "Neutral," "Satisfied," and "Very Satisfied". This scale allows patients to express their level of satisfaction with various aspects of their surgical experience.
  Very Dissatisfied/Very Unsatisfied (1): Indicates a very negative experience. Dissatisfied/Unsatisfied (2): Indicates a negative experience. Neutral (3): Indicates neither satisfaction nor dissatisfaction. Satisfied (4): Indicates a positive experience. Very Satisfied (5): Indicates a very positive experience.
Pain Visual Analog Scale (Pain - VAS) Score | Baseline and 3, 6, 12, and 24 months
  a measurement tool used to gauge subjective experiences, especially pain, by having individuals mark a spot on a continuous line between two defined extremes, representing, for example, "no pain" and "worst pain".
Lachmeter | Baseline and Months 3, 6, 12, and 24
  A Lachmeter is a device that is attached above and below your knee, that will measure the laxity (looseness) of your knee.
Lachman pivot shift | Baseline and 3, 6, 12, and 24 months
  The Lachman, pivot shift tests are all physical examination techniques used to assess the integrity of the anterior cruciate ligament (ACL) in the knee.
Lachman anterior drawer | Baseline and 3, 6, 12, and 24 months
  The Lachman anterior drawer tests are all physical examination techniques used to assess the integrity of the anterior cruciate ligament (ACL) in the knee.
Tegner Activity Score | Baseline and 3, 6, 12, and 24 months
  The Tegner Activity Scale (TAS) is a simple, self-administered questionnaire that assesses a patient's level of activity, both at work and in sports, on a scale of 0 to 10The TAS is a 1-item questionnaire scored on a scale of 0 to 10.
  0: represents maximum disability due to knee problems, such as being on sick leave or disability.
  10: represents participation in competitive sports at a national or international elite level, like soccer.
Time to Return to Sport/Previous Activity Level | Months 3, 6, 12, and 24
  Time to Return to Sport/Previous Activity Level
Y-Balance Distance | Months 6, 12, and 24
  asked to reach a maximum distance in 3 different directions (shape of a "Y") - do this while standing on 1 leg and staying balanced. Both legs will be tested
Number of Single Hop | Months 6, 12, and 24
  asked to perform a maximum single leg broad jump - 2 reps on each leg
Number of Triple Hops | Months 6, 12, and 24
  asked to perform a single leg triple hop (hop forward 3 times in a row) - 2 reps on each leg
Biodex Strength Testing | Months 6, 12, and 24
  measure the strength of your thigh muscles (quadriceps and hamstrings) - kick leg forward and pull leg backward as hard as possible - perform this assessment at 1 to 2 different speeds (the machine controls the speed). Both legs will be tested.
Reoperation Rate | Months 3, 6, 12, and 24
  Reoperation Rate
Failure Rate | Months 3, 6, 12, and 24
  Failure Rate
Brace Compliance Rate | Months 6, 12, and 24
  While wearing the brace, the sensor will track how many hours the brace is in use. The goal of the sensor is to track compliance of wearing the brace during rehabilitative and sport (or military) specific activity.
Number of Brace Complications | Months 6, 12, and 24
  Number of Brace Complications

CONTACTS AND LOCATIONS:
Overall Officials: Brian Waterman, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No